CLINICAL TRIAL: NCT03860831
Title: Lecturer of Anesthesia ,Intensive Care and Pain Management in Faculty of Medicine Ain Shams University
Brief Title: Intranasal Ketamine and Midazolam Mixture for Procedural Sedation in Children With Mental Disabilities:
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Sanaa Farag Mahmoud Wasfy, lecturer of aneathesia, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: R 57/2018
Record Dates: First submitted 2018-11-12; First posted 2019-03-04 (Actual); Last update posted 2019-03-08 (Actual); Status verified 2019-03

CONDITIONS: Procedural Sedation
Keywords: nasal; sedation; developmental delay
MeSH Terms: conditions — Learning Disabilities | interventions — Ketamine; Midazolam

STUDY DESIGN:
Intervention Model Description: 2 groups of children aged 4-12 years with mental disabilities(autism,down syndrome,cerebral palsy)
Who Masked: Care Provider, Outcomes Assessor
Masking Description: surgeon who are providing medical procedure and nurse who records vital data and level of sedation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intranasal (IN) (Experimental): Group IN will receive nasal ketamine+midazolam mixture by mucosal atomisation device: midazolam (0.2 mg/kg) +ketamine (5mg/kg).
  the calculated dose will be equally divided into the two nostrils by the parents
  Interventions: Drug: Ketamine + midazolam
- intramuscular (IM) (Active Comparator): Group IM will receive intramuscular administration of liquid ketamine +midazolam mixture:midazolam (0.2 mg/kg) +ketamine (5mg/kg) in the gluteal region.
  Mild to moderate restraint was done with the help of the parents during drug administration.
  Interventions: Drug: Ketamine + midazolam

INTERVENTIONS:
Drug: Ketamine + midazolam — Group IN received intranasal midazolam (0.2 mg/kg) +ketamine (5mg/kg). Group IM received intramuscular midazolam (0.2 mg/kg) +ketamine (5mg/kg) in the gluteal region.
  Other Names: ketalar +dormicum

SUMMARY:
Ketamine and Midazolam are well known sedative drugs that can be given through different routes such as intravenous, intramuscular, oral, rectal and intranasal route. Anesthetic staff usually prefer intravenous route but sometimes inserting venous access is difficult in uncooperative mentally disabled children. Intranasal ketamine+Midazolam can be a needless effective alternative in these vulnerable patients

DETAILED DESCRIPTION:
Sedation and analgesia decreases the need for general anesthesia outside the operating room. Intravenous route is the standard way of sedation, but its use can be limited in uncooperative mentally disabled children. Active Physical restraint of children causes emotional trauma for both parents and children particularly in these patients. Oral sedation has multiple disadvantages as delayed onset of action, better taste, the need of different types of syrup or honey according to the preference of the patient, children may refuse to take oral drugs or even spit it and it also causes postoperative nausea and vomiting. In contrast, intramuscular sedation is an easy effective way of administration and it is preferred due to its rapid onset of action and higher predictability of the duration, however, fear of the pain of injections is considered a disadvantage in this vulnerable pediatric patients. nasal route is an important alternative route because it is a painless and needless approach with rapid drug absorption from nasal mucosa reaching the cerebrospinal fluid and bypassing the first pass metabolism in the liver. Intranasal midazolam for sedation of children was first described by Wilton et al .Recently studies proved the use of nasal ketamine spray for treatment of resistant depression in adults. Ketamine as a premedication in children has been also successfully given through the nasal route. In Ain shams University hospitals we give either oral Midazolam or intramuscular Ketamine followed by sevoflurane or propofol for pediatric procedural sedation. Nasal Midazolam or Ketamine has not been tried despite being a feasible choice with many possible advantages. Combination of ketamine and midazolam causes deeper sedation and less dysphoric reaction of ketamine so in this study, we evaluate the efficacy and safety of administration of this combination through intranasal route for procedural sedation in children with mental developmental delay outside the operating room.

After approval from our Ethical Committee, written informed consent from the parents will be taken. Forty children presented with autism,mongolism or cerebral palsy classified as American Society of Anesthesiologists (ASA) physical status I and II, aged between 4 and 12 years will be enrolled in our study, and computer-generated assignment will be used for randomization and to allocate patients to one of two equal study groups.

patients will fulfill the fasting hours if elective while the patients in ER will be asked to wait for six hours after last meal.

Patients will be divided into two groups Group IN:will receive intranasal ketamine 5 mg/kg and midazolam 0.2 mg/kg, and we will give intranasal sedatives by using mucosal atomisation device.

Group IM:will receive intramuscular ketamine 5 mg/kg, and midazolam 0.2 mg/kg Sedation levels after 10, 20, and 30 min will be evaluated by Pediatric Sedation State Scale (PSSS).

Drugs will be given 15- 20 minutes before procedure then Heart rate (HR), Oxygen saturation (Spo2), and mean arterial blood pressure (MBP) will be continuously monitored and recorded every 5 min after drug administration for 60 minutes .

Local anesthesia will be given in painful procedures. Intravenous ketamine 1 mg/kg will be given if needed due to prolongation of procedure or if required sedation level not reached through intranasal or intramuscular route.

respiratory events as airway obstruction and desaturation less than 92% will be treated by jaw thrust and oxygen supplementation, apnea or laryngeal spasm will be managed with endotracheal intubation. Wheezing will be recorded and properly managed with bronchodilators and steroids.

Emergency cart and drugs will be available for haemodynamic and respiratory instabilities.

After recovery of the patients, parents and doctors will rate their overall satisfaction by using simple image of 5 point Likert scale.

Primary outcome: effectiveness of sedation. Secondary outcome: onset, duration of sedation, adverse effect, parents and doctor satisfaction.

End point of the study: if our technique failed to sedate the patients general anesthesia will be given either intravenous ketamine 1mg/kg or inhalational sevoflurane to complete the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria of the patients were:
* Mentally affected children (autism,down syndrome and cerebral palsy)
* children who are scheduled for Short procedures (30 minutes or less) under sedation

Exclusion Criteria:

* parents refusal.
* child cooperation and acceptance of venipuncture or cannula in situ.
* children with known allergy to ketamine or midazolam.
* liver or renal organ dysfunction.
* suspected difficult cannulation.
* congenital heart disease.
* active pulmonary infection or asthma.
* increased intracranial tension or intraocular pressure.
* severe trauma0
* significant nasal discharge or obstruction.

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2019-03-06 (Actual); Primary Completion 2019-06 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
change in sedation level after intranasal or intramuscular ketamine midazolam mixture administration. | every 10 minutes through the study till one hour after administration
  sedation level measured by Pediatric Sedation State Scale (PSSS): State 5: Movement impedes procedure and requires forceful immobilization
  State 4: Movement requires gentle immobilization for positioning
  State 3: Facial expression of pain or anxiety
  State 2: Quiet, not moving, no frown, no verbalization of complaint (ideal state)
  State 1: Deeply asleep with normal vital signs, but requires airway intervention or assistance (e.g., central or obstructive apnea)
  State 0: Deeply asleep with abnormal physiologic parameters that require acute intervention (e.g., O2 saturation <90%, hypotension, bradycardia)
  highest score is 0 and least score is 5

SECONDARY OUTCOMES:
parents satisfaction | two hours after administration
  image form of 5 point likert scale. 5-very satisfied 4-Satisfied 3-Neither satisfied nor dissatisfied 2-Dissatisfied
  1-Very dissatisfied least score is 1 and highest score is 5

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Sanaa Farag Mahmoud, Cairo, New Cairo
  - Ainshams hospitals, Cairo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Malamed SF. Sedation: A Guide to Patient Management. New York, NY: CV: Mosby-Year Book Inc; 1995. 3rd ed.
- [Background] Lee-Kim SJ, Fadavi S, Punwani I, Koerber A. Nasal versus oral midazolam sedation for pediatric dental patients. J Dent Child (Chic). 2004 May-Aug;71(2):126-30. PMID 15587094
- [Background] Ochs-Ross R,et al. Efficacy and safety of intranasal esketamine plus an oral antidepressant in eldely patients with treatment-resistant depression.Poster PS066 presented at CINP 2018,16-19 june, Vienna, Austria.
- [Background] Dallimore D, Herd DW, Short T, Anderson BJ. Dosing ketamine for pediatric procedural sedation in the emergency department. Pediatr Emerg Care. 2008 Aug;24(8):529-33. doi: 10.1097/PEC.0b013e318180fdb5. PMID 18645539
- [Background] Cravero JP, Askins N, Sriswasdi P, Tsze DS, Zurakowski D, Sinnott S. Validation of the Pediatric Sedation State Scale. Pediatrics. 2017 May;139(5):e20162897. doi: 10.1542/peds.2016-2897. PMID 28557732